CLINICAL TRIAL: NCT00671060
Title: Misoprostol for Treatment of Fetal Death at 14-28 Weeks of Pregnancy, Inclusive, Not Accompanied by Complete Expulsion of the Contents of the Uterus
Brief Title: Misoprostol for Treatment of Fetal Death at 14-28 Weeks of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Stanford University (Other); Albert Einstein College of Medicine (Other); University of Florida (Other); Huong Vuong Hospital (Unknown); Boston Medical Center (Other); Christiana Care Health Services (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3.3; 1R01FD003107-01A1 (FDA)
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Intrauterine Fetal Demise
Keywords: intrauterine fetal death; misoprostol
MeSH Terms: conditions — Stillbirth | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Women in Group 1 will be administered two tablets (2 100 mcg misoprostol tablets), which she will be instructed to hold in her cheeks for 200 minutes, after which she will swallow any medication that remains. In cases where cervical dilation is not complete after six hours, women will be given a second dose of study drug. Study drug will continue to be administered at 6-hourly intervals through hour 42 after the study dose.
  Interventions: Drug: Misoprostol
- 1 (Placebo Comparator): Women in Group 1 will be administered two tablets (a 100 mcg misoprostol tablet and a placebo tablet made to resemble a 100 mcg misoprostol tablet), which she will be instructed to hold in her cheeks for 200 minutes, after which she will swallow any medication that remains. In cases where cervical dilation is not complete after six hours, women will be given a second dose of study drug. Study drug will continue to be administered at 6-hourly intervals through hour 42 after the study dose.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 200 mcg buccal misoprostol administered every 6 hours for up to 48 hours until fetus is delivered.
  Arms: 2
Drug: Misoprostol — 100 mcg buccal misoprostol administered every 6 hours for upto 48 hours
  Arms: 1

SUMMARY:
The purpose of the proposed study is to test - in a randomized, blinded trial - two different doses of the prostaglandin E1 analogue misoprostol administered buccally as a treatment for fetal death at 14 - 28 weeks, inclusive, of pregnancy. At such an advanced stage of pregnancy, the nonviable fetus is often not spontaneously evacuated, and yet timely evacuation is vital in order to avoid the possibility of, among other things, potentially life-threatening maternal coagulopathies. Current approaches to uterine evacuation in these cases include dilatation and evacuation (D&E) surgery (in less advanced pregnancies) and labor induction with a variety of products. Misoprostol has been demonstrated to be as effective as, or more effective than, either oxytocin or prostaglandin E2 analogues for this indication in a number of small, non-FDA-approved trials which have been published in the peer-reviewed literature. In the absence of more formal study of this treatment, however, dosages are not standardized, pathways of administration vary, and other uncertainties linger. The purpose of the protocol proposed herein is to formally establish, via a randomized, double-blinded study, the safety and effectiveness of misoprostol for this indication, and to compare the value of two distinct doses, so that providers may henceforward proceed with greater authority and confidence.

ELIGIBILITY:
Inclusion Criteria:

* Women presents with spontaneous fetal death
* Gestational age of fetus between 14-28 weeks

Exclusion Criteria:

* Transmural uterine scar;
* Allergies or other contraindications to use of misoprostol;
* Placental abruption with active hemorrhage;
* Complete placenta previa;
* Extreme uterine structural anomalies;
* Or other contraindications to vaginal delivery of the fetus;
* Presentation in active labor (moderate to severe contractions every 10 minutes); or
* Four or more previous deliveries

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (5):
- United States (4):
  - Stanford University, Palo Alto, California
  - Christiana Care Health System, Newark, Delaware
  - University of Illinois at Chicago, Chicago, Illinois
  - Albert Einstein College of Medicine, The Bronx, New York
- Huong Vuong Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- See also: Related Info — http://www.gynuity.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized trial was conducted at Montefiore Medical Center, Stanford University, Stroger Hospital, Christiana Care Hospital, the Huong Vuong Hospital in Ho Chi Minh City, Viet Nam. Women who sought medical care for possible fetal demise in pregnancies of between 14 and 28 weeks from December 2008 to December 2011 were screened.
Pre-assignment Details: No participants were excluded from the trial before assignment to groups.
Groups:
- 200 Mcg: Women in Group 1 will be administered two tablets (2 100 mcg misoprostol tablets), which she will be instructed to hold in her cheeks for 200 minutes, after which she will swallow any medication that remains. In cases where cervical dilation is not complete after six hours, women will be given a second dose of study drug. Study drug will continue to be administered at 6-hourly intervals through hour 42 after the study dose.
- 100 Mcg: Women in Group 1 will be administered two tablets (a 100 mcg misoprostol tablet and a placebo tablet made to resemble a 100 mcg misoprostol tablet), which she will be instructed to hold in her cheeks for 200 minutes, after which she will swallow any medication that remains. In cases where cervical dilation is not complete after six hours, women will be given a second dose of study drug. Study drug will continue to be administered at 6-hourly intervals through hour 42 after the study dose.
Period: Overall Study
Arm/Group | 200 Mcg | 100 Mcg
Started | 77 | 76
Completed | 76 (1 woman completed study but was excluded from analysis because gestational age <14 weeks.) | 75 (1 woman was withdrawn from the study due to preeclampsia.)
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 Mcg | 100 Mcg | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 73 | 73 | 146
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.6 (5.6) | 25.8 (5.9) | 25.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 76 | 153
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
  Vietnam | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Successful Expulsion of Fetus and Placenta Within 48 Hours
Time Frame: 48 hours
Population: One woman assigned to the 200μg arm was determined to be ineligible after enrollment due to a gestational age less than 14 weeks. She was not included in the analysis. One woman in the 100mcg arm was withdrawn from the study due to preeclampsia. She was included in the analysis as a failed induction.
Measure: Number; unit: participants
Arm/Group | 200 Mcg | 100 Mcg
Number analyzed (Participants) | 76 | 76
participants | 60 | 47
Statistical Analysis 1: Comparison: 200 Mcg vs 100 Mcg; Rates of success were compared across study arms. The study was a separate, non-comparative efficacy study. In order to have 80% power (alpha=.05) to demonstrate that each misoprostol regimen was 95%, ± 5%, effective, we enrolled 73 women in each arm of the study, or 146 women total. The sample size also provided 80% power (alpha=.05) to detect a significant difference between treatments should 200μg prove 98% effective and 100μg prove 88% effective; Test type: Superiority or Other; p < 0.05, Chi-squared; Risk Ratio (RR) = 0.682

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | 200 Mcg | 100 Mcg
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/76
Other Adverse Events (participants affected / at risk) | 1/77 | 0/76
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 Mcg (N=77) | 100 Mcg (N=76)
Other adverse event (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other